CLINICAL TRIAL: NCT05221879
Title: Anti-factor Xa Based Venous Thromboembolism Prophylaxis: Dose Adjustment in ICU Patients
Brief Title: Anti-factor Xa Based Venous Thromboembolism Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MMC-18-0262
Record Dates: First submitted 2022-01-09; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Dose Adjustment of Enoxaparin in ICU Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with target factor 10a levels (No Intervention): Patients with target factor 10a levels continued to recieve the standard Enoxaparin dose of 40 mg SC daily.
- Patients with sub-therapuetic factor 10a levels (Other): In patients with sub-therapuetic factor 10a levels we increased the Enoxaparin dose to 60 mg SC daily.
  Interventions: Other: Dose adjustment of Enoxaparin in patients with sub-therapuetic (prophylactic) levels of factor 10a

INTERVENTIONS:
Other: Dose adjustment of Enoxaparin in patients with sub-therapuetic (prophylactic) levels of factor 10a — We screened ICU patients who recieved DVT prophylaxis with fixed dose of Enoxaparin (40 mg SC daily) for peak blood levels of factor 10A. For patients who did not achieve therapuetic 10a levels (0.2-0.4) we increased the Enoxaparin dose to 60 mg SC daily.
  Arms: Patients with sub-therapuetic factor 10a levels

SUMMARY:
Introduction: Venous thromboembolism (VTE) in the intensive care unit (ICU) is associated with significant morbidity and mortality therefore prevention is imperative to reduce its burden. VTE prophylaxis in ICU patients is primarily pharmacological using low molecular weight heparin. This study aims to determine the proportion of ICU patients receiving VTE prophylaxis that achieves appropriate anti-factor Xa activity (aFXa) prophylactic levels and to characterize this patient population Methods: Seventy-five patients admitted to the General ICU were included. Peak and trough aFXa levels were measured at 4 and 23 hours respectively after receiving the second consecutive daily enoxaparin 40 mg sc injection. Patients in whom peak aFXa levels were found to be sub-prophylactic, peak and trough levels were repeated as above

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria were age over 18 years and a predicted ICU stay of more than 72 h.

-

Exclusion Criteria: Exclusion criteria were any contraindication for heparin-based thromboembolic prophylaxis, patients with an indication for therapeutic anticoagulation , administration of unfractioned-heparin or low-molecular-weight-heparin prior to study entry, active hemorrhage, or creatinine clearance < 30 mL/min.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-06-23 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Peak aFXa levels following 2 consecutive doses of sc 40 mg enoxaparin | Up to 72 hours from ICU admission.
  We measured peak aFXa levels following 2 consecutive doses of sc 40 mg enoxaparin among ICU patients who recieved enoxaparin for VTE prophylaxis..

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No